CLINICAL TRIAL: NCT02672150
Title: Juvenile Justice Translational Research on Interventions for Adolescents in the Legal System: Multi-site Implementation Study
Brief Title: Juvenile Justice Translational Research on Interventions for Adolescents in the Legal System
Acronym: (JJ-TRAILS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Columbia University (Other); Emory University (Other); Mississippi State University (Other); Temple University (Other); Texas Christian University (Other); University of Kentucky (Other)
Responsible Party: Principal Investigator, Michael L. Dennis, Ph.D., Coordinating Center Multi-PI, Chestnut Health Systems
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: JJ-TRIALS; U01DA036221 (NIH); U01DA036226 (NIH); U01DA036233 (NIH); U01DA036176 (NIH); U01DA036225 (NIH); U01DA036224 (NIH); U01DA036158 (NIH)
Record Dates: First submitted 2016-01-22; First posted 2016-02-03 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Substance Use Disorders
Keywords: evidence-based practice implementation; system change; interagency collaboration; substance use; treatment services; data-driven decision making; juvenile justice; adolescents; justice-involved youth; cluster randomized trial
MeSH Terms: conditions — Substance-Related Disorders | interventions — GAT

STUDY DESIGN:
Intervention Model Description: Staff from 34 juvenile community supervision agencies were observed for a 6 month baseline period than trained over 4 months on using a behavioral health service cascade model to screen, identify, and refer youth to substance use treatment. Half the sites were randomized to 12 additional months of facilitation. Sites were then monitored for an additional 4 month maintenance phase.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Pairs of sites were optimally randomize based on 10,000 trials to the two conditions by the coordinating center. The assignment (to core or core+enhanced) was not revealed to the local research center or site until after completion of the core. Thus it is double blind.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): During the Baseline Control data is collected in all 36 sites at the agency, staff, and youth level on the 6 months prior to the interventions in Arms 2 & 3 to document what practice was before the study.
- Core (Active Comparator): In the second phase (after baseline) all 36 sites receive a Core condition that includes five interventions: (1) JJ-TRIALS Orientation Meetings, (2) Needs Assessment, (3) Behavioral Health Training, (4) Site Feedback Report, (5) Goal Achievement Training, (6) Monthly Site Check-ins, and (7) Quarterly Reports. As part of Goal Achievement Training, sites receive assistance in using their Site Feedback Reports to select goals to meet their local needs. Sites are trained on using Data-Driven Decision Making (DDDM) to inform decisions (e.g., selecting a goal, monitoring progress) and enlisting DDDM templates and tools (developed as part of the project) to plan and implement proposed changes.
  these principles to their improvement efforts during the implementation phase.
  Interventions: Behavioral: Core
- Enhanced (Experimental): While the core intervention and DDDM are expected to facilitate change, organizations may need additional support to apply these principles to their improvement efforts during the implementation phase. In the third phase (after Core), 1/2 of the sites are randomly assigned to an Enhanced condition that provides continuing support for the use of DDDM tools by adding research staff facilitation of DDDM over a 12-month period and formalized Local Change Teams (LCTs) featuring representation from the JJ agency and a local BH provider, with meetings facilitated by research staff).
  Interventions: Behavioral: Core; Behavioral: Enhanced

INTERVENTIONS:
Behavioral: Core
  Other Names: GAT, DDDM
  Arms: Core; Enhanced
Behavioral: Enhanced
  Other Names: DDDM, Facilitation
  Arms: Enhanced

SUMMARY:
This is a multi site experiment to evaluate the impact of various strategies for increasing the use of evidence based screening, assessment and linkage to substance use treatment. All sites collect baseline data and receive a core intervention. Half are then randomly assigned to get an additional year of coaching to facilitate implementation.

DETAILED DESCRIPTION:
Background: The Juvenile Justice-Translational Research on Interventions for Adolescents in the Legal System (JJ-TRIALS) study is a cooperative implementation science initiative involving the National Institute on Drug Abuse, six Research Centers, a Coordinating Center, and Juvenile Justice Partners representing seven U.S. states. The pooling of resources across Centers enables a robust implementation study design involving 36 juvenile justice agencies and their behavioral health partner agencies, coproducing a study protocol that has potential to advance implementation science, meets the needs of all constituencies (funding agency, researchers, partners, study sites), and can be implemented with fidelity across the cooperative can be challenging.

Methods/design: The JJ-TRIALS primary study uses a head-to-head cluster randomized trial with a phased rollout to evaluate the differential effectiveness of two conditions (Core and Enhanced) in 36 sites located in 7 states. Core strategies for promoting change are compared to an Enhanced strategy that incorporate all core strategies plus active facilitation. Target outcomes include improvements in evidence-based screening, assessment, and linkage to substance use treatment.

Primary Research Questions:

1. Does the Core and/or Enhanced Intervention reduce unmet need by increasing Cascade retention related to screening, assessment, treatment initiation, engagement and continuing care?
2. Does the addition of the Enhanced Intervention components further increase the percentage of youth retained in the Cascade relative to the Core components?
3. Does the addition of the Enhanced Intervention components improve service quality relative to Core sites?
4. Do staff perceptions of the value of best practices increase over time, and are increases more pronounced in Enhanced sites?

ELIGIBILITY:
Specific site inclusion criteria include: (a) ability to provide youth service records, (b) service to youth under community supervision, (c) access to treatment provider(s) if treatment is not provided directly by the JJ agency, (d) participation in requisite intervention training/activities,(e) minimum average case flow of 10 youth per month, (f) minimum of 10 staff per site, and (g) a senior JJ staff member who agrees to serve as site leader/liaison during the study. Study sites are geographically dispersed and were identified by state JJ agencies (and not selected for particular substance use or related BH service needs).

Youth inclusion criteria include: all youth entering the juvenile justice system during the period within the exception of those who are already in treatment at the time that they are referred to the juvenile justice agency.

Staff inclusion criteria include: all staff actively working with the youth under community supervision in the site with exclusion only of higher level administrative or regional staff over multiple units..

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 839 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Service Cascade: % Referred to Substance Use Treatment | 120 weeks
  Calculated from juvenile justice and substance use treatment agency records as the number of youth referred to substance use treatment divided by the number of youth identified as need of substance use treatment.
Staff Perception: Value of Evidenced Based Substance Use Treatment | 120 weeks
  Calculated from staff surveys at juvenile justice and substance use treatment agencies as the average staff ranking of the perceived "value" of using of evidence-based substance use treatment services.

SECONDARY OUTCOMES:
Service Cascade: % Screened for Substance Use Problems | 120 weeks
  Calculated from juvenile justice and substance use treatment agency records as the number of youth "Screened" for substance use problems divided by the number of youth entering the juvenile justice system.
Service Cascade: % Clinically Assessed for Substance Use Problems | 120 weeks
  Calculated from juvenile justice and substance use treatment agency records as the number of youth "Clinically Assessed" for substance use problems divided by the number of youth entering the juvenile justice system.
Service Cascade: % In Need of Substance Use Treatment | 120 weeks
  Calculated from juvenile justice and substance use treatment agency records as the number of youth identified (via screening, clinical assessment or other sources) as "In Need of Substance Use Treatment" divided by the number of youth entering the juvenile justice system.
Service Cascade: % Initiating Substance Use Treatment | 120 weeks
  Calculated from juvenile justice and substance use treatment agency records as the number of youth "Initiating" Substance Use Treatment within 90 days of referral" divided by the number referred to treatment from the juvenile justice system.
Service Cascade: % Engaged in Substance Use Treatment | 120 weeks
  Calculated from juvenile justice and substance use treatment agency records as the number of youth "Engaged" in Substance Use Treatment for 6 weeks or more weeks divided by the number initiating treatment.
Service Cascade: % With Substance Use Treatment Continuing Care | 120 weeks
  number of youth "Continuing" to receive substance use treatment services forCalculated from juvenile justice and substance use treatment agency records as the 90 days or more divided by the number initiating treatment.
Service Quality: Timing of Screening or Clinical Assessment | 120 weeks
  Calculated from juvenile justice and substance use treatment agency records as the mean days from entry into the justice system to the first of screening or clinical assessment for substance use problems.
Service Quality: Timing of Substance Use Treatment Initiation | 120 weeks
  Calculated from juvenile justice and substance use treatment agency records as the mean days from referral to and initiation of substance use treatment.
Service Quality: Number of Evidence Based Practices | 120 Weeks
  Based on agency surveys and youth records from juvenile justice and substance use treatment agencies, the number of steps using 1 or more evidenced based practices in each of the following steps along the service cascade: screening, clinical assessment, referral, substance use treatment.
Staff Perception: Value of Evidenced Based Screening | 120 weeks
  Calculated from staff surveys at juvenile justice and substance use treatment agencies as the average staff ranking of the perceived "value" of using of evidence-based screening.
Staff Perception: Value of Evidenced Based Clinical Assessment | 120 weeks
  Calculated from staff surveys at juvenile justice and substance use treatment agencies as the average staff ranking of the perceived "value" of using of evidence-based clinical assessment.
Staff Perception: Value of Evidenced Based Substance Use Prevention | 120 weeks
  Calculated from staff surveys at juvenile justice and substance use treatment agencies as the average staff ranking of the perceived "value" of using of evidence-based substance use prevention.
Staff Perception: Value of Evidenced Based HIV Risk Prevention | 120 weeks
  Calculated from staff surveys at juvenile justice and substance use treatment agencies as the average staff ranking of the perceived "value" of using of evidence-based HIV Risk prevention.

CONTACTS AND LOCATIONS:
Overall Officials: Tisha R Wiley, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA); Gail A Wasserman, Ph.D., Principal Investigator — Columbia University; Ralph DiClemente, Ph.D., Principal Investigator — Emory University; Gene H Brody, Ph.D., Principal Investigator — Emory University; Angela A Robertson, Ph.D., Principal Investigator — Mississippi State University; Steven R Belenko, Ph.D., Principal Investigator — Temple University; Danica K Knight, Ph.D., Principal Investigator — Texas Christian University; Carl G Leukefeld, Ph.D., Principal Investigator — University of Kentucky; Michael L Dennis, Ph.D., Principal Investigator — Chestnut Health Systems; Christy K Scott, Ph.D., Principal Investigator — Chestnut Health Systems
Locations (8):
- United States (8):
  - Emory University, Atlanta, Georgia
  - Chestnut Health Systems, Bloomington, Illinois
  - University of Kentucky, Lexington, Kentucky
  - National Institute on Drug Abuse, Rockville, Maryland
  - Mississippi State University, Starkville, Mississippi
  - Columbia University, New York, New York
  - Temple University, Philadelphia, Pennsylvania
  - Texas Christian University, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
The coordinating center is charged with creating de-identified versions of agency, staff and client level service data available at the end of the study.

REFERENCES:
- [Derived] Jones SD, Bartkowski JP, Belenko S, Becan JE, Taxman FS, Wasserman GA, Aarons GA, McReynolds LS, Dolbear C, Xu X. Site engagement in implementation research: Introducing SEAMLIS as a conceptual and measurement framework. Health Justice. 2025 Jul 5;13(1):44. doi: 10.1186/s40352-025-00349-1. PMID 40616691
- [Derived] Nelson V, Wood J, Belenko S, Pankow J, Piper K. Conditions of successful treatment referral practices with justice-involved youth: Qualitative insights from probation and service provider staff involved in JJ-TRIALS. J Subst Use Addict Treat. 2024 Jul;162:209358. doi: 10.1016/j.josat.2024.209358. Epub 2024 Mar 27. PMID 38548060
- [Derived] Belenko S, Dembo R, Knight DK, Elkington KS, Wasserman GA, Robertson AA, Welsh WN, Schmeidler J, Joe GW, Wiley T. Using structured implementation interventions to improve referral to substance use treatment among justice-involved youth: Findings from a multisite cluster randomized trial. J Subst Abuse Treat. 2022 Sep;140:108829. doi: 10.1016/j.jsat.2022.108829. Epub 2022 Jun 19. PMID 35751945
- [Derived] Marks KR, Leukefeld CG, Dennis ML, Scott CK, Funk R; JJ-TRIALS Cooperative. Geographic differences in substance use screening for justice-involved youth. J Subst Abuse Treat. 2019 Jul;102:40-46. doi: 10.1016/j.jsat.2019.04.005. Epub 2019 Apr 13. PMID 31202287
- [Derived] Fisher JH, Becan JE, Harris PW, Nager A, Baird-Thomas C, Hogue A, Bartkowski JP, Wiley T; JJ-TRIALS Cooperative. Using Goal Achievement Training in juvenile justice settings to improve substance use services for youth on community supervision. Health Justice. 2018 Apr 30;6(1):10. doi: 10.1186/s40352-018-0067-4. PMID 29713840
- [Derived] Becan JE, Bartkowski JP, Knight DK, Wiley TRA, DiClemente R, Ducharme L, Welsh WN, Bowser D, McCollister K, Hiller M, Spaulding AC, Flynn PM, Swartzendruber A, Dickson MF, Fisher JH, Aarons GA. A model for rigorously applying the Exploration, Preparation, Implementation, Sustainment (EPIS) framework in the design and measurement of a large scale collaborative multi-site study. Health Justice. 2018 Apr 13;6(1):9. doi: 10.1186/s40352-018-0068-3. PMID 29654518
- [Derived] Belenko S, Knight D, Wasserman GA, Dennis ML, Wiley T, Taxman FS, Oser C, Dembo R, Robertson AA, Sales J. The Juvenile Justice Behavioral Health Services Cascade: A new framework for measuring unmet substance use treatment services needs among adolescent offenders. J Subst Abuse Treat. 2017 Mar;74:80-91. doi: 10.1016/j.jsat.2016.12.012. Epub 2016 Dec 31. PMID 28132705
- [Derived] Knight DK, Belenko S, Wiley T, Robertson AA, Arrigona N, Dennis M, Bartkowski JP, McReynolds LS, Becan JE, Knudsen HK, Wasserman GA, Rose E, DiClemente R, Leukefeld C; JJ-TRIALS Cooperative. Juvenile Justice-Translational Research on Interventions for Adolescents in the Legal System (JJ-TRIALS): a cluster randomized trial targeting system-wide improvement in substance use services. Implement Sci. 2016 Apr 29;11:57. doi: 10.1186/s13012-016-0423-5. PMID 27130175
- See also: JJTRIALS home page — http://www.nida.nih.gov/jjtrials